CLINICAL TRIAL: NCT01856621
Title: Pharmacokinetic Study Comparing Two Salmeterol Fluticasone Propionate Device-metered Dry Powder Inhalers, Salmeterol/Fluticasone Easyhaler and Seretide Diskus 50/500 Mcg/Inhalation; a Randomised, Doubleblind,Single Centre, Single Dose, Crossover Study in Healthy Subjects
Brief Title: Comparison of Salmeterol and Fluticasone Propionate Absorption From Salmeterol/Fluticasone Easyhaler With Seretide Diskus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 3106008 EudraCT 2012-003782-18
Record Dates: First submitted 2013-05-15; First posted 2013-05-17 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Charcoal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Seretide Diskus and charcoal (Active Comparator): Single-dose of Seretide Diskus (50/500 mcg/inhalation) and charcoal
  Interventions: Drug: Seretide Diskus and charcoal
- Seretide Diskus (Active Comparator): Single-dose of Seretide Diskus (50/500 mcg/inhalation)
  Interventions: Drug: Seretide Diskus
- SF Easyhaler and charcoal (Experimental): Salmeterol/fluticasone Easyhaler (50/500 mcg/inhalation) with charcoal
  Interventions: Drug: SF Easyhaler and charcoal
- SF Easyhaler (Experimental): Salmeterol/fluticasone Easyhaler (50/500 mcg/inhalation)
  Interventions: Drug: SF Easyhaler

INTERVENTIONS:
Drug: Seretide Diskus and charcoal — 2 inhalations as a single dose
  Arms: Seretide Diskus and charcoal
Drug: Seretide Diskus — 2 inhalations as a single dose
  Arms: Seretide Diskus
Drug: SF Easyhaler and charcoal — 2 inhalations as a single dose
  Arms: SF Easyhaler and charcoal
Drug: SF Easyhaler — 2 inhalations as a single dose
  Arms: SF Easyhaler

SUMMARY:
The purpose of this study is to compare the test product Salmeterol/fluticasone Easyhaler with the reference product Seretide Diskus in terms of drug absorbed in the bloodstream.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females aged 18-60 years
* Normal weight, at least 50 kg

Exclusion Criteria:

* Evidence of clinically significant cardiovascular, renal, hepatic, haematological, GI, pulmonary, metabolic-endocrine, neurological or psychiatric disease
* Any clinically significant abnormal laboratory value or physical finding that may interfere with the interpretation of study results or constitute a health risk for the subject if he/she takes part in the study
* Any condition requiring regular concomitant treatment (including vitamins and herbal products) or likely to need any concomitant treatment during the study
* Known hypersensitivity to the active substance(s) or the excipient of the drug
* Pregnant or lactating females

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter Cmax of plasma salmeterol concentration | Within 34 h
Pharmacokinetic parameter Cmax of plasma fluticasone propionate concentration | Within 34 h
Pharmacokinetic parameter AUCt of plasma salmeterol concentration | Within 34 h
Pharmacokinetic parameter AUCt of plasma fluticasone propionate concentration | Within 34 h

CONTACTS AND LOCATIONS:
Locations (1):
- Orion Pharma Clinical Pharmacology Unit, Espoo, Finland